CLINICAL TRIAL: NCT06827002
Title: Cissus Quadrangularis (CQR-300®) and Dichrostachys Glomerata (Dyglomera®) Extracts Increase GLP-1 Levels and Inhibit Dipeptidyl Phosphate-4 Activity in Healthy Overweight and Obese Adults
Brief Title: Effect of Aqueous Extracts of Cissus Quadrangularis and Dichrostachys Glomerata on GLP-1 Concentration and DPP-4 Activity in Overweight and Obese Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Yaounde 1 (Other)
Collaborators: J & A Oben Foundation (Unknown)
Responsible Party: Principal Investigator, Pr. Julius Oben, Head of Department, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JAOFCissusDyglo; JAOF122025 (Other Grant/Funding Number: J & A Oben Foundation); N°2014/08/488/CE/CNERSH/SP (Other: National Ethics Committee of Cameroon); BTC-JIRB2023-084 (Other: University of Yaounde I IRB)
Record Dates: First submitted 2025-01-29; First posted 2025-02-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Obesity and Overweight; Appetite Regulation
Keywords: Natural Products; GLP-1; DDP-4 Inhibitors; Obesity management; Appetite regulation; CQR-300®; Dyglomera®
MeSH Terms: conditions — Obesity; Overweight | interventions — Dextrins; semaglutide

STUDY DESIGN:
Intervention Model Description: The study involves Two hundred and forty eight (248) overweight or obese participants (25 ≥ BMI ≤ 34), randomly divided into four groups: the placebo, DGE group, CQE and semaglutide groups.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo Group (Placebo Comparator): 62 participants aged 18-65 with a BMI between 25 - 34 kg/m 2 randomly assigned to the placebo group will be administered a 400 mg dextrin capsule daily for 12 weeks. Participants will be instructed to maintain their usual lifestyle and dietary habits and to report any delays in taking the capsules.
  Interventions: Drug: Dextrin
- Dichrostachys glomerata Extract (DGE) Group (Experimental): 62 participants aged 18-65 with a BMI between 25 - 34 kg/m 2 randomly assigned to the DGE group will be administered 400mg DGE capsule daily for 12 weeks. Participants will be instructed to maintain their usual lifestyle and dietary habits and to report any delays in taking the capsules.
  Interventions: Drug: Dichrostachys glomerata
- Cissus quadrangularia Extract (CQE) Group (Experimental): 62 participants aged 18-65 with a BMI between 25 - 30 kg/m 2 randomly assigned to the CQE group will be administered 300mg CQE capsule daily for 12 weeks. Participants will be instructed to maintain their usual lifestyle and dietary habits and to report any delays in taking the capsules.
  Interventions: Drug: Cissus quadrangularia
- Semaglutide Group (Active Comparator): 62 participants aged 18-65 with a BMI between 25 - 34 kg/m 2 randomly assigned to the semaglutide group will be administered a repackaged Oral semaglutide (Rybelsus®) capsule daily (4-week dose escalation from 3 to 7 to 14mg). Participants will be instructed to maintain their usual lifestyle and dietary habits and to report any delays in taking the capsules.
  Interventions: Drug: Semaglutide (Rybelsus®)

INTERVENTIONS:
Drug: Dichrostachys glomerata — DGE were procured from Gateway Health Alliances, Fairfield in 400 mg and 300 mg capsules.
  Other Names: Dyglomera®; DGE
  Arms: Dichrostachys glomerata Extract (DGE) Group
Drug: Cissus quadrangularia — CQR-300® were procured from Gateway Health Alliances, Fairfield in 400 mg and 300 mg capsules.
  Other Names: CQR-300®; CQE
  Arms: Cissus quadrangularia Extract (CQE) Group
Drug: Dextrin — Placebo capsules containing 400 mg of dextrin, looking identical to DGE and CQE were also procured from Gateway Health Alliances, Fairfield, California, USA.
  Other Names: Placebo group
  Arms: Placebo Group
Drug: Semaglutide (Rybelsus®) — Oral semaglutide (Rybelsus®) was purchased and then repackaged into capsules looking identical to DGE, CQE and placebo capsules.
  Other Names: semaglutide
  Arms: Semaglutide Group

SUMMARY:
Obesity is a global health crisis affecting over 2.3 billion individuals worldwide. This prospective study aims to evaluate the comparative effects of standardised Cissus quadrangularis extract (CQE) and Dichrostachys glomerata extract (DGE) on obesity-related parameters, focusing on their impact on glucagon-like peptide-1 (GLP-1) levels and dipeptidyl peptidase-4 (DPP-4) enzyme activity in obese subjects. Parameters such as GLP-1 levels, DPP-4 activity, food intake, satiety, body weight, blood lipids, fasting blood glucose, and visceral fat mass will be measured at baseline and various intervals.

In our previous pre-clinical trial involving 18 adult male Wistar rats (150-200 g), randomly divided into three groups: a control group fed a normal diet, and two treatment groups receiving DGE (400 mg/kg) or CQE (300 mg/kg) alongside a normal diet, the results demonstrated that both DGE and CQE significantly increased GLP-1 levels and inhibited DPP-4 activity compared to the control group. These effects were associated with reduced food intake, body weight, and fasting blood glucose levels. Additionally, both extracts positively modified blood lipid profiles, with significant changes in HDL, LDL, and triglyceride levels. The findings suggest that DGE and CQE exert their anti-obesity effects through mechanisms involving GLP-1 enhancement and DPP-4 inhibition, offering potential therapeutic pathways for weight management and metabolic health.

This prospective study aims to provide clinical evidence supporting the use of these plant extracts in addressing obesity and its related complications.

DETAILED DESCRIPTION:
Obesity is a health burden affecting over 2.3 billion people of all ages globally. The development and progression of obesity involve a complex pathogenesis, and several drugs have been developed to target these pathways. In recent years, dipeptidyl peptidase-4 (DPP-4) inhibitors or gliptins, such as sitagliptin, saxagliptin, and vildagliptin, have been considered as a viable obesity management option. Gliptins inhibit DPP-4, an enzyme known to deactivate the GLP-1 hormone, contributing to the development and progression of obesity and other metabolic diseases. GLP-1 is one of the important incretin hormones secreted in the L-cells of the gut for the maintenance of blood sugar homeostasis. It exhibits other pleiotropic effects through its receptors in the liver, brain, and stomach to delay gastric emptying, reduce appetite, and induce significant weight loss. In healthy individuals, GLP-1 has a half-life of >2 minutes due to the activities of DPP-4 . Some studies have observed higher DPP-4 levels in obese individuals, further reducing the incretin effects of GLP-1. Gliptins are primarily invented to manage type 2 diabetes. However, their weight loss effects are quite significant, presenting as a potent management option for obesity.

Synthetically produced drugs are often associated with side effects and contraindications. For conditions such as obesity, patients often require unique management options due to sensitivity and the high likelihood of comorbidities. For instance, obese individuals are more vulnerable to pancreatitis and pancreatic cancer, whereas gliptins are associated with a high incidence of acute pancreatitis. Gliptins also present other side effects such as upper respiratory infections, headache, urinary tract infections, arthralgia, and in severe cases, Stevens-Johnson syndrome. Cost-wise, gliptins are considerably expensive. The current FDA-approved gliptins are intended for the management of diabetes. Prescribing them for obesity may lead to higher demand and prices as well as scarcity. Hence, there is a need for a wider range of safe, cost-effective, and potent alternatives.

Natural products continue to emerge as potential drug leads for several metabolic disease conditions due to their potency and low toxicity. DGE (Dichrostachys glomerata), a popular Cameroonian spice, and CQE (Cissus quadrangularis), an ornamental and medicinal plant growing in Africa and Asia, have shown tremendous effects on weight loss. A recent study showed that DGE induced 22.85% weight loss in 60 subjects in 12 weeks. In a double-blind placebo-controlled study involving 35 subjects, CQE reduced body fat by 12.8% in 8 weeks. The mechanism of these two extracts is not fully understood. It has been proposed that DGE and CQE are anorectic. Some studies suggested that DGE and CQE reduced food intake through increased adiponectin secretion and the AMPK pathway.

Additionally, CQE was shown to boost serotonin levels. Serotonin has received much attention in weight loss research in the past. It has been implicated for its appetite-suppressing effect on the arcuate nucleus hypothalamus, a region responsible for food intake and energy expenditure.

Up to the present, no study has investigated the effect of DGE or CQE on GLP-1 or DPP-4 levels. Hence, this study aims to evaluate the efficacy of DGE and CQE as potent alternatives to gliptins in obesity management.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant/non-lactating females
* Participants aged 18 to 65 years old
* Participants with BMI between 25 and 34 kg/m²
* Participants willing to comply with the study protocol

Exclusion Criteria:

* Participants younger than 18 years or older than 65 years
* Participants not available for the study period
* Morbid obesity (BMI > 34.9 kg/m²)
* Diabetes mellitus requiring daily insulin management
* Pregnancy or breastfeeding
* Active infection
* Systemic diseases, including HIV/AIDS, Active hepatitis, Clinical signs of active malignancy within the past 5 years
* Use of any medication or natural health product that might affect the parameters of interest in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Dyglomera® and CQR-300® on participants GLP-1 level | Baseline (Week 0), Week 4, Week 8, and Week 12
  Description: GLP-1 levels will be determined in pg/mL using the RayBio® GLP-1 ELISA kit.
Effect of Dyglomera® and CQR-300® on participants BMI | Baseline (Week 0), Week 4, Week 8, and Week 12
  BMI will then be calculated as follows:
  BMI (kg/m²)=Weight in Kg/Height in meter²
Effect of Dyglomera® and CQR-300® on participants Fasting blood glucose | Baseline (Week 0), Week 4, Week 8, and Week 12
  Glucose levels will be measured in blood samples taken from each participant after a 12-hour fast at baseline (Week 0), Week 4, Week 8, and Week 12 using the glucose oxidase-peroxidase enzymatic method with a OneTouch Ultra 2 glucometer.
  Unit of measure: mg/dL
Effect of Dyglomera® and CQR-300® on participants DPP4 activity | Baseline (Week 0), Week 4, Week 8, and Week 12
  DPP-4 activity will be measured using Cayman's DPP-4 inhibitor screening assay kit according to the manufacturer's instructions.
  Unit of Measure: % Activity Remaining
  This will be determined using the calculation below:
  % activity remaining = (slope of test sample/positive control slope) × 100.
Effect of Dyglomera® and CQR-300® on participants Lipid Profile | Baseline (Week 0), Week 4, Week 8, and Week 12
  Blood lipid levels (cholesterol, triglycerides, and HDL-c) will be measured in blood samples taken from each participant after a 12-hour fast at baseline (Week 0), Week 4, Week 8, and Week 12 using ChronoLab commercial kits according to the protocol of the manufacturers. LDL-c will be assessed using the Friedewald et al. formula.
  LDL-c = Plasma-c - HDL-c - Total Plasma triglyceride/5 Unit of measure: mg/dL
Effect of Dyglomera® and CQR-300® on participants Body Fat percentage | Baseline (Week 0), Week 4, Week 8, and Week 12
  The body fat percentage (%) was measured using an impedance meter at visits 1, 2 (week 0 or baseline), 3 (week 4), 4 (week 8), and 5 (week 12).
Effect of Dyglomera® and CQR-300® on participants Body weight | Baseline (Week 0), Week 4, Week 8, and Week 12
  Body weight will be measured in Kg using a TANITA brand scale at Visits 1, 2 (Week 0/Baseline), 3 (Week 4), 4 (Week 8), and 5 (Week 12).

SECONDARY OUTCOMES:
Effect of Dyglomera® and CQR-300® on participants' energy Intake | Week 12
  Participants will maintain a food diary for seven consecutive days (the last week of each study period), recording all foods, drinks, and snacks consumed. Food intake will be recorded in household measurements and converted into grams using manufacturer labels where applicable. Nutrient intake (carbohydrates, lipids, and proteins) will then be quantified in grams using the FAO food composition table for Cameroon.
  Energy intake will be calculated as follows:
  EI (Kcal/day) = ECarb + ELip + EProt
  where: ECarb(Kcal/day)=Amount of carb ingested (g) x 4 Kcal/7 Eprot (Kcal/day)=Amount of carb/prot ingested (g) x 4 Kcal/7 ELip (Kcal/day)=Amount of lipid ingested (g) x 9 Kcal/7
  Considering that: 1 g carbohydrate or protein = 4 Kcal and 1 g lipid = 9 kcal

CONTACTS AND LOCATIONS:
Overall Officials: Julius E Oben, PhD, Principal Investigator — University of Yaounde 1
Locations (1):
- University of Yaounde 1, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
* Metabolic parameters (Blood sugar, Blood lipid),
  * Anthroprmetric measures (height, weight, BMI and body fat percentage)
  * DPP-4 and GLP-1 levels data collected through out the study

REFERENCES:
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Youovop J, Takuissu G, Mbopda C, Nwang F, Ntentié R, Mbong M, Azantsa B, Singh H, Oben J. The effects of Dyglomera® (Dichrostachys glomerata extract) on body fat percentage and body weight: a randomized, double-blind, placebo-controlled clinical trial. Functional Foods in Health and Disease 2023, 13: 334-346.
- [Background] Filipova EP, Uzunova KH, Vekov TY. Comparative analysis of therapeutic efficiency and costs (experience in Bulgaria) of oral antidiabetic therapies based on glitazones and gliptins. Diabetol Metab Syndr. 2015 Jul 16;7:63. doi: 10.1186/s13098-015-0059-7. eCollection 2015. PMID 26288659
- [Background] Filippatos TD, Panagiotopoulou TV, Elisaf MS. Adverse Effects of GLP-1 Receptor Agonists. Rev Diabet Stud. 2014 Fall-Winter;11(3-4):202-30. doi: 10.1900/RDS.2014.11.202. Epub 2015 Feb 10. PMID 26177483
- [Background] Tkac I, Raz I. Combined Analysis of Three Large Interventional Trials With Gliptins Indicates Increased Incidence of Acute Pancreatitis in Patients With Type 2 Diabetes. Diabetes Care. 2017 Feb;40(2):284-286. doi: 10.2337/dc15-1707. Epub 2016 Sep 22. PMID 27659407
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Valerio CM, de Almeida JS, Moreira RO, Aguiar LBS, Siciliano PO, Carvalho DP, Godoy-Matos AF. Dipeptidyl peptidase-4 levels are increased and partially related to body fat distribution in patients with familial partial lipodystrophy type 2. Diabetol Metab Syndr. 2017 Apr 24;9:26. doi: 10.1186/s13098-017-0226-0. eCollection 2017. PMID 28450900
- [Background] Ahren B, Schmitz O. GLP-1 receptor agonists and DPP-4 inhibitors in the treatment of type 2 diabetes. Horm Metab Res. 2004 Nov-Dec;36(11-12):867-76. doi: 10.1055/s-2004-826178. PMID 15655721
- [Background] van Bloemendaal L, Ten Kulve JS, la Fleur SE, Ijzerman RG, Diamant M. Effects of glucagon-like peptide 1 on appetite and body weight: focus on the CNS. J Endocrinol. 2014 Mar 7;221(1):T1-16. doi: 10.1530/JOE-13-0414. Print 2014 Apr. PMID 24323912
- See also: WHO. Obesity and Overweight. — https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT06827002/Prot_SAP_000.pdf